CLINICAL TRIAL: NCT01600989
Title: Mitochondrial Function of Immune Cells in Severe Sepsis and Septic Shock - a Prospective Observational Cohort Study
Brief Title: Mitochondrial Function of Immune Cells in Sepsis
Acronym: MitoSepsis
Status: Completed | Type: Observational
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Other Study IDs: 015/10
Record Dates: First submitted 2012-05-11; First posted 2012-05-17 (Estimated); Last update posted 2014-04-25 (Estimated); Status verified 2014-04

CONDITIONS: Shock, Septic
Keywords: shock septic; monocytes; lymphocytes; mitochondria; interleukins; Tumor Necrosis Factor-alpha; Hypoxia-Inducible Factor 1, alpha Subunit
MeSH Terms: conditions — Shock, Septic | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum, isolated B-cells, T-cells, Monocytes
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Patients with severe sepsis / septic shock: 30 Adult patients (age > 18years), with severe sepsis or septic shock as defined by the 2001 SCCM/ESICM/ACCP/ATS/SIS International Sepsis Definitions Conference guidelines at the time of admission to ICU.
  Interventions: Other: blood sampling
- Healthy volunteers: Healthy volunteers
  Interventions: Other: blood sampling

INTERVENTIONS:
Other: blood sampling — Blood samples will be taken at ICU admission, and 24h and 48h after admission, and at time of resolution of sepsis
  Groups: Patients with severe sepsis / septic shock
Other: blood sampling — Blood samples will be taken twice at a 7 day interval
  Groups: Healthy volunteers

SUMMARY:
Introduction: Evidence suggests that sepsis and septic shock severely impair mitochondria and that the resulting mitochondrial dysfunction is related to the severity and outcome of the resulting organ dysfunction. In sepsis mitochondrial abnormalities - biochemical and ultrastructural - have been recognized in multiple organs, including liver, kidney, skeletal and heart muscle tissue and blood cells. Circulating immune cells play an important role in the pathophysiology of sepsis. Stimulation of the immune system alters the energy requirements of immune cells; down-regulation of immune-cell activity has been associated with prolonged sepsis and unfavourable outcome. The aim of the project is to comprehensively investigate changes in mitochondrial function of immune cells in patients with severe sepsis and septic shock. The following main hypotheses will be evaluated:

* Severe sepsis and septic shock leads to increased energy requirements of immune cells and to an increase in mitochondrial enzyme activities and energy production.
* Changes of mitochondrial function in human immune cells are associated with alterations in clinical and laboratory markers of severity of sepsis.
* Prolonged sepsis and unfavourable outcome is associated with down regulation of mitochondrial function.

Methods: A total of 30 adult patients admitted to the intensive care unit (ICU) due to severe sepsis or septic shock will be included in the study; 30 healthy volunteers serve as controls. Patients with any type of chronic infectious, inflammatory or autoimmune diseases, after transplantations or receiving immunosuppressive agents are excluded.

Collected baseline characteristics include patient demographics, diagnosis and severity of illness scores at the time of admission. Daily collected follow up data include clinical and laboratory parameters of organ dysfunction, use of vasopressors/inotropes, use of antibiotics, use of steroids and results of microbiological cultures/stains.

Negative identification and isolation of monocytes, B cells and CD4 T cells will be performed daily from ICU admission to discharge using an antibody-antigen mediated immunomagnetic cell isolation procedure that depletes all blood cells except the specific target cells. Mitochondrial function of immune cells will be assessed by measurement of mitochondrial complex activity for complexes I to IV by a standard titration protocol. Additionally, the levels of pro- and anti-inflammatory cytokines (Interleukin (IL)-1, IL-6, IL-10, TNF-α) will be assessed throughout the stay in the ICU. For comparison mitochondrial function of of monocytes, B cells and CD4 T cells and cytokine levels will be measured in a group of 10 healthy volunteers.

Analysis plan: Changes in mitochondrial function of immune cells over time compared to a healthy control group and during the course of severe sepsis and septic shock is the main outcome parameter of this study. Assessed predictors are determined by the severity of the underlying septic condition and include clinical and laboratory evidence for dysfunction of vital organ systems and changes in levels of inflammatory and anti-inflammatory cytokines.

DETAILED DESCRIPTION:
Background

Evidence suggests that sepsis and septic shock severely impair mitochondria and that the resulting mitochondrial dysfunction is related to the severity and outcome of the resulting organ dysfunction. In sepsis mitochondrial abnormalities - biochemical and ultrastructural - have been recognized in multiple organs, including liver, kidney, skeletal and heart muscle tissue and blood cells. A systematic review on mitochondrial function assessed as oxygen consumption, state 3 and state 4 respiration, respiratory enzyme activity, or tissue ATP levels and turnover rates showed decreased function especially in sepsis models lasting more than 16h . Depleted levels of reduced glutathione, an important intra-mitochondrial antioxidant, in combination with increased generation of reactive oxygen species (ROS) and reactive nitrogen species (RNS) inhibit oxidative phosphorylation and ATP generation. This acquired intrinsic derangement in cellular energy metabolism contributes to reduced activities of mitochondrial electron transport chain enzyme complexes and impaired ATP biosynthesis and contributes to the organ dysfunction in sepsis.

Circulating immune cells play an important role in the pathophysiology of sepsis. Stimulation of the immune system alters the energy requirements of immune cells; down-regulation of immune-cell activity has been associated with prolonged sepsis. Immune cell activation mandates an increase in energy requirements, thus a reduced production of ATP due to impaired mitochondrial function may be a factor in modulating the immune response in sepsis. Alterations in mitochondrial function and energetic failure have been reported in peripheral blood mononuclear cells and seem to be associated with the modulation of the immune response to sepsis. Macrophages incubated with endotoxin/interferon-γ show a decrease in oxygen consumption and inhibition of mitochondrial I complex. Different mechanisms for alteration of mitochondrial function in these cells have been proposed, including increases in NO production and nitration of mitochondrial proteins [14], elevation of IL-10 [15] or prostaglandin levels. In human neutrophils intact mitochondrial function plays an important role in chemotaxis and phagocytosis, impairment of these mechanisms leads to a decreased defence ability to microbial challenges.

HIF-1α is a transcription factor that acts as a key regulatory factor in the evolution of oxygen homeostasis. Under normoxic conditions HIF-1α is continuously synthesized and degraded after hydroxylation by dioxygenases that utilize oxygen, Fe and α-ketoglutarate as substrates. During hypoxia, the low availability of oxygen limits the reaction; HIF-1α is no longer degraded and rapidly accumulates and triggers the transcription of genes involved in oxygen homeostasis such as glycolytic enzymes, glucose transporters, vascular endothelial growth factor (VEGF) and erythropoietin. Under hypoxic conditions, HIF mediates also a decrease in mRNA levels of the respiratory chain proteins, preparing the cell to produce ATP mainly from glycolysis and not from oxidative phosphorylation, thereby optimizing cell energetics and homeostasis for survival and function during hypoxia.

Recent published reports have linked inflammation and endotoxin stimulation to HIF-1α activation. HIF-1α has been shown to be up-regulated and stabilized in LPS-treated macrophages and monocytes under normoxic conditions. HIF-1α levels were shown to be decreased in macrophages deficient in TLR4 after LPS stimulation, suggesting that LPS stimulation of HIF-1α is mediated by TLR4.

Data on mitochondrial function of human immune cells in severe sepsis is limited and the potential correlation of mitochondrial energy requirements and production and the severity of the patient's condition and outcome are not well established. The immunologic reaction in the context of severe sepsis and septic shock consists of an interdependent, highly complex system that involves different types of immune cells and pro- and anti-inflammatory cytokines involved in a time-dependent process. Simple in-vitro studies assessing mitochondrial function of a single type of immune cells and single cytokines just a one point in time during the course of the septic process might not be an appropriate model to mirror the complex interactions of the immune system. Serial measurements of mitochondrial function of different key-player cells and specific pro- and anti-inflammatory cytokines and apoptosis markers parallel with other clinical and laboratory markers of sepsis may offer a more in-depth evaluation and understanding of this deleterious disease pattern.

Objective

The aim of the project is to comprehensively investigate changes in mitochondrial function and morphology of immune cells in patients with severe sepsis and septic shock. We plan to assess changes in mitochondrial function of monocytes, B cells and CD4+ T cells in correlation to levels of various cytokines and to classic clinical and laboratory parameters of severity of sepsis and outcome.

Methods

A total of 30 patients admitted to the intensive care unit (ICU) of a tertiary care hospital due to severe sepsis or septic shock will be included in the study after obtaining written informed consent of the patient or the patient's next of kin. Patients with any type of chronic infectious, inflammatory or autoimmune diseases, after transplantations or receiving immunosuppressive agents are excluded.

Controls: 30 healthy volunteers Assessment of mitochondrial function of monocytes/granulocytes will be performed by measurement of mitochondrial complex activity using a standard titration protocol to measure activation of complex I to IV. To measure serum levels of IL-1, IL-6, IL-10 and TNF standard commercial kits will be used.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (age > 18years)
* Severe sepsis or septic shock as defined by the 2001 SCCM/ESICM/ACCP/ATS/SIS International Sepsis Definitions Conference guidelines at the time of admission to ICU.

Exclusion Criteria

* Patients with any type of chronic infectious, inflammatory or autoimmune diseases
* Patients after hematopoietic or solid organ transplantation
* Patients receiving long term treatment with steroids or other immunosuppressive agents

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 30 patients with severe sepsis or septic shock at ICU admission
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2012-05; Primary Completion 2013-10 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Mitochondrial function of immune cells | At the time of ICU admission

SECONDARY OUTCOMES:
Change from baseline in mitochondrial function of immune cells | 24 hours after ICU admission
Change from baseline in mitochondrial function of immune cells | 48 hours after ICU admission
Change from baseline in mitochondrial function of immune cells | At time of resoltion of sepsis, expected to be after 5 days
Levels of cytokines (of IL-1, IL-6, IL-10 and TNFa) | At ICU admission, 24h and 48h after admission, & at time of resolution of sepsis (expected to be after 5 days)
ICU mortality | At time of dismissal from ICU, expected to be after 7 days

CONTACTS AND LOCATIONS:
Overall Officials: Tobias Merz, Study Chair — Department of Intensive Care Medicine, Bern University Hospital (Inselspital) and University of Bern
Locations (1):
- Department of Intensive Care Medicine, Bern University Hospital (Inselspital) and University of Bern, Bern, Switzerland